CLINICAL TRIAL: NCT00739219
Title: Management of Asthma Patients Guided by Exhaled Nitric Oxide (eNO) Using the Apieron NO Analyzer
Brief Title: Management of Asthma Patients Guided by Exhaled Nitric Oxide (eNO)
Acronym: Outcomes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated due to lack of care guidelines in the protocol.
Sponsor: Apieron (Industry)
Responsible Party: Nina Peled, VP of Regulatory and Clinical Affairs, Apieron
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP00006
Record Dates: First submitted 2008-08-19; First posted 2008-08-21 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2008-10

CONDITIONS: Asthma
Keywords: Asthma; inflammation; nitric oxide; eNO; FENO
MeSH Terms: conditions — Asthma; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- eNO group (Active Comparator): eNO measurement is used to inform asthma management decisions
  Interventions: Device: Apieron Insight eNO monitor
- control group (No Intervention): Asthma is managed according to existing standard of care

INTERVENTIONS:
Device: Apieron Insight eNO monitor — The Apieron Insight(tm) eNO monitor is used to measure exhaled nitric oxide, and asthma is managed to keep eNO below an individualized target.
  Arms: eNO group

SUMMARY:
This study is designed to show that pharmacotherapy guided by eNO and clinical standard of care produces a superior outcome to trial-based therapy guided by clinical standard of care alone.

DETAILED DESCRIPTION:
Patients with persistent, moderate to severe asthma will be randomized to receive therapy guided by either eNO and clinical standard of care (eNO group) or clinical standard of care (control group). An eNO treatment algorithm will be established for each patient in the eNO group at Baseline (Visit 1). Enrollment is estimated to be six months with a follow up period of twelve months.

ELIGIBILITY:
Inclusion Criteria:

* Pre-existing diagnosis of asthma
* Persistent, moderate or severe asthma as classified by NAEPP
* Sub-optimally controlled asthma
* Initiated ICS therapy for at least the past 30 days and a history of improvement of asthma control on steroids

Exclusion Criteria:

* Active cigarette smoking or ≥ 10 pack-years smoking history
* Xolair taken in the past 6 months prior to enrollment
* Oral prednisone taken in the last 4 weeks prior to enrollment
* Cystic Fibrosis, COPD, ciliary dyskinesia, chest wall deformities or scoliosis
* Subject is currently enrolled in another investigational drug study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2006-12; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Asthma control days | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: William E Berger, MD, MBA, Principal Investigator — Southern California Research
Locations (12):
- United States (12):
  - Southern California Research, Mission Viejo, California
  - Allergy & Asthma Associates of Santa Clara Valley Research Center, San Jose, California
  - Allergy Associates of Hartford, Glastonbury, Connecticut
  - Asthma and Allergy Center of Chicago, S.C., River Forest, Illinois
  - The Asthma- Allergy Clinic& Research Center, Shreveport, Louisiana
  - Chesapeake Clinical Research, Baltimore, Maryland
  - The Clinical Research Center, LLC, St Louis, Missouri
  - Center for Allergy and Asthma, Highland Park, New Jersey
  - Pulmonary & Allergy Associates P.A., Summit, New Jersey
  - Allergy, Asthma & Dermatology Research Center, LLC, Lake Oswego, Oregon
  - Asthma & Allergy Research Associates, Upland, Pennsylvania
  - Pharmaceutical Research & Consulting, Inc., Dallas, Texas